CLINICAL TRIAL: NCT06610799
Title: Phase Ib Study to Evaluate the Safety, Tolerability and Efficacy of IBI363 in Combination with Oxaliplatin and Capecitabine (XELOX) in First-line Treatment of Unresectable Advanced or Metastatic Gastric and Gastroesophageal Junction Adenocarcinoma
Brief Title: Study of IBI363 in Patients with Advanced First-line Gastric Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xiangdong Cheng (Other)
Responsible Party: Sponsor-Investigator, Xiangdong Cheng, Secretary of the party committee, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI363Y110
Record Dates: First submitted 2024-09-18; First posted 2024-09-24 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-09

CONDITIONS: IBI363 + Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cohort 1 (Experimental): IBI363 combination with oxaliplatin and capecitabine (XELOX) for first-line treatment of unresectable advanced or metastatic gastric and gastroesophageal junction adenocarcinoma
  Interventions: Drug: IBI363

INTERVENTIONS:
Drug: IBI363 — IBI363 Q3W Oxaliplatin 130 mg/m2，IV，Q3W, Capecitabine ,1000mg/ m2，PO，Bid，d1-14，Q3W

SUMMARY:
This is a phase 1b study designed to evaluate the safety, tolerability and efficacy of IBI363 in combination with oxaliplatin and capecitabine (XELOX) in first-line treatment of unresectable advanced or metastatic gastric and gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, ≥ 18 years and ≤75 years.
2. Subjects with unresectable advanced or metastatic gastric and gastroesophageal junction adenocarcinoma without prior systematic treatment.
3. Subjects with at least one measurable lesion according to RECIST v1.1.
4. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1.
5. Expected survival time ≥ 3 months.

Exclusion Criteria:

1. Women who are pregnant or lactating, or intending to become pregnant before, during, or within 6 months after the last dose of study drug.
2. Active uncontrolled bleeding or a known bleeding diathesis.
3. Subjects with history of or known active seizure disorder, brain metastases, spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Through out the study (up to 2 years)
  The efficacy of solid tumors was evaluated according to RECIST v1.1
Disease control rate (DCR) | Through out the study (up to 2 years)
  The efficacy of solid tumors was evaluated according to RECIST v1.1

SECONDARY OUTCOMES:
Progression Free Survival（PFS）; | Up to 2 years
  The efficacy of solid tumors was evaluated according to RECIST v1.1
Overall Survival, OS） | Up to 2 years
  The efficacy of solid tumors was evaluated according to RECIST v1.1
Adverse Enent (AE), Treatment-Emergent AE (TEAE), Adverse Event of Special Interest (AESI) and Serious Adverse Event (SAE) | Up to 90 days after the last administration
  Adverse events will be assessed by investigator(s) according to NCI-CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided